CLINICAL TRIAL: NCT03102463
Title: The Role of Milk Derived Peptides on Glycaemic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: Enterprise Ireland (Other Government)
Responsible Party: Principal Investigator, Prof Helen M Roche, Associate Professor, University College Dublin
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: FHI-3
Record Dates: First submitted 2016-02-26; First posted 2017-04-05 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Insulin Resistance
Keywords: Insulin sensitivity; Obesity; Insulin resistance; Milk derived hydrolysate; Hyperinsulinemic-euglycaemic clamp
MeSH Terms: conditions — Insulin Resistance; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Water Control (Sham Comparator)
  Interventions: Dietary Supplement: Water Control; Other: Lipid Load
- Milk derived hydrolysate (Active Comparator)
  Interventions: Dietary Supplement: Milk derived hydrolysate; Other: Lipid Load
- Parent Protein (Active Comparator)
  Interventions: Dietary Supplement: Parent Protein; Other: Lipid Load

INTERVENTIONS:
Dietary Supplement: Water Control — 120mL water given as a control, followed by a hyperinsulinemic-euglycaemic clamp
  Arms: Water Control
Dietary Supplement: Milk derived hydrolysate — Milk derived hydrolysate made up as a milkshake in 120mL water, followed by a hyperinsulinemic-euglycaemic clamp
  Arms: Milk derived hydrolysate
Dietary Supplement: Parent Protein — Parent protein made up as a milkshake in 120mL water, followed by a hyperinsulinemic-euglycaemic clamp
  Arms: Parent Protein
Other: Lipid Load — 100mL oral lipid load

SUMMARY:
This study aims to ascertain the potential of novel milk derived hydrolysates to improve glycaemic control to promote metabolic health. A comprehensive characterisation of the metabolic response to these milk derived hydrolysates will ascertain the effect of the hydrolysates in terms of insulin sensitivity. These hydrolysates have been shown to improve insulin resistance in cell and animal models. Therefore the investigators aim is to test their efficacy in overweight, insulin resistant individuals at risk of developing type 2 diabetes.

DETAILED DESCRIPTION:
Recent figures estimate 60% of Irish adults are overweight or obese. As obesity is associated with the development of insulin resistance, which precedes type 2 diabetes development by decades, novel food based solutions are required to improve glycaemic control and attenuate insulin resistance.

In the current study insulin resistant individuals will undergo 4 study visits, 1 screening visit and 3 subsequent visits. At each of the 3 visits they will receive an oral lipid load consisting of 100mL soya bean oil, followed by either a water control; the hydrolysate being tested or the parent protein from which the hydrolysate was derived. After which they will undergo a 4 hour hyperinsulinemic-euglycaemic clamp at each visit to assess their insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65 years
* BMI > 26 kg/m2
* Prepared to maintain a constant body weight for the duration of the study
* Free of any chronic or infectious disease
* Not taking any medication for the regulation of blood sugars
* Diet controlled type 2 diabetes
* Free of any milk allergies or lactose intolerance
* Without anaemia

Exclusion Criteria:

* <18 or >65 years
* Diabetes (pharmacologically treated) or other endocrine disorders.
* Chronic inflammatory conditions.
* Kidney or liver dysfunction.
* Anaemia (Haemoglobin <12g/dl men, < 11g/dl women).
* Taking any medication for the regulation of blood sugars.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-10; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Glucose Disposal Rate | 12 weeks
  M-value (mg/kg/min) /Glucose disposal rate will be used to measure of insulin sensitivity

SECONDARY OUTCOMES:
Markers of glycaemic control | 12 weeks
  Glucose (mmol/L)
Markers of glycaemic control | 12 weeks
  Insulin (mU/L)inflammatory markers
Lipid Profile | 12 weeks
  Non-esterified fatty acids (mmol/L)
Lipid Profile | 12 weeks
  Triglycerides (mmol/L) and other related lipid markers
Inflammatory Markers | 12 weeks
  High sensitivity C reactive protein (mg/L)
Inflammatory Markers | 12 weeks
  C-peptide (ng/mL) and other related

CONTACTS AND LOCATIONS:
Overall Officials: Helen M Roche, PhD, Principal Investigator — University College Dublin
Locations (1):
- St Vincent's University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No